CLINICAL TRIAL: NCT06124339
Title: Interventions to Promote Brain Health Virtual Reality Study
Brief Title: Brain Health Virtual Reality Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Judy Pa, Co-Director of ADCS, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 803273
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Aging; Aging Problems; Memory Loss; Memory Impairment; Memory Disorders in Old Age; Memory Disorder, Spatial; Memory Disorders; Mild Cognitive Impairment; Cognitive Decline; Cognitive Change; Cognition Disorders in Old Age
Keywords: Virtual Reality; technology; intervention; exercise; cycling; memory; brain health; aging
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Motor Activity | interventions — Exercise; Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive activity - VR spatial navigation only (Active Comparator): VR spatial navigation program will consist of a spatial navigation program that increases difficulty and length per trial over time. Spatial navigation is the ability to navigate between multiple elements/landmarks widely used in computer games. A trial is a test of performance or quality of someone or something.
  Interventions: Behavioral: Cognitive Activity (VR)
- Physical activity - Cycling only (Active Comparator): The physical activity program will consist of a stationary bike cycling program. Each day will consist of a cycling program of varying levels of difficulty for 20-50 minutes.
  Interventions: Behavioral: Physical Activity
- Combined, simultaneous physical and cognitive activity (Experimental): The combined physical and cognitive activity VR program will consist of a spatial navigation program that increases difficulty and length per trial over time.
  Interventions: Behavioral: Physical and Cognitive Activity

INTERVENTIONS:
Behavioral: Physical Activity — There will be three sessions a week over the course of 16 weeks.
  Arms: Physical activity - Cycling only
Behavioral: Cognitive Activity (VR) — There will be three sessions a week over the course of 16 weeks.
  Arms: Cognitive activity - VR spatial navigation only
Behavioral: Physical and Cognitive Activity — There will be three sessions a week over the course of 16 weeks.
  Arms: Combined, simultaneous physical and cognitive activity

SUMMARY:
The Interventions for Brain Health Virtual Reality Study is a NIH-funded clinical research trial at the University of California San Diego (UCSD) Health under the supervision of the study principal investigator Dr. Judy Pa. The overarching goal of this trial is to use a novel virtual reality (VR) based intervention that simultaneously engages physical and cognitive activity aimed at improving brain health and cognition in older adults. The investigators will compare 3 types of interventions: physical activity, VR cognitive activity, and combined VR physical and cognitive activity over 16 weeks to evaluate physical and brain health changes.

ELIGIBILITY:
Inclusion Criteria:

1. 50-85 years of age
2. Fluent in English
3. Can safely ride a stationary bike

Exclusion Criteria:

1. Dementia
2. History of a neurological disorder
3. Severe sensory deficits
4. Inability to perform intervention (e.g., inability to cycle safely)
5. Contraindications to MRI scan (e.g., pacemaker)
6. Fear of needles/ blood
7. Prior history of fainting due to sight of needles of blood

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2028-08-08 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
MST memory performance | 16 Weeks
  With the study's primary focus on hippocampal function, we will use the Mnemonic Separation Task (MST), a hippocampus-dependent discrimination test of similar objects, as our primary cognitive outcome. The MST is a memory task designed to heavily tax memory processes for making fine discriminations between highly similar objects or unrelated objects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes